CLINICAL TRIAL: NCT03382821
Title: A Prospective Randomized Comparative Trial of Targeted Injection Via a Transforaminal Approach With Dexamethasone Versus an Epidural Catheter Via an Interlaminar Approach With Particulate Steroid for the Treatment of Cervical Radicular Pain
Brief Title: Comparative Trial Via Tranforaminal Approach Versus Epidural Catheter Via Interlaminar Approach
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Epimed (Industry)
Responsible Party: Principal Investigator, Zack McCormick, Zachary L. McCormick, MD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 105766
Record Dates: First submitted 2017-12-04; First posted 2017-12-26 (Actual); Results first posted 2021-03-22 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Cervical Radiculopathy
Keywords: cervical epidural steroid injection; transforaminal approach; epidural catheter targeted; interlaminar approach; cervical radicular pain
MeSH Terms: conditions — Radiculopathy | interventions — Dexamethasone; Triamcinolone; dexamethasone 21-phosphate; Lidocaine; Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, comparative trial
Who Masked: Participant
Masking Description: Each subject will be randomized into a group assignment in a 1:1 manner, #1 or #2, as outlined in the Methods section
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Transforaminal ESI with dexamethasone (Active Comparator): Group 1: Transforaminal cervical ESI with dexamethasone sodium phosphate
  Interventions: Procedure: Transforaminal ESI with dexamethasone; Drug: Dexamethasone Sodium Phosphate 10 MG/ML; Drug: Lidocaine
- Transforaminal catheter-targeted ESI with triamcinolone (Active Comparator): Group 2: Catheter-targeted cervical ESI with triamcinolone acetonide
  Interventions: Procedure: Transforaminal catheter-targeted ESI with triamcinolone; Drug: Lidocaine; Drug: Triamcinolone Acetonide 40mg/mL

INTERVENTIONS:
Procedure: Transforaminal ESI with dexamethasone — Catheter-targeted ESI via interlaminar access at the C7-T1 level with dexamethasone sodium phosphate 1.5 mL (10 mg/mL) and 1 ml 1% lidocaine (total volume 2.5 mL).
  Arms: Transforaminal ESI with dexamethasone
Procedure: Transforaminal catheter-targeted ESI with triamcinolone — Catheter-targeted ESI via interlaminar access at the C7-T1 level with triamcinolone acetonide 2 mL (40mg/mL) and 1 ml 1% lidocaine (total volume 3 mL).
  Arms: Transforaminal catheter-targeted ESI with triamcinolone
Drug: Dexamethasone Sodium Phosphate 10 MG/ML — Transforaminal ESI with dexamethasone 1.5 mL of dexamethasone sodium phosphate in group #1
  Arms: Transforaminal ESI with dexamethasone
Drug: Lidocaine — 1 mL of 1% lidocaine as diluent for the steroid in both group #1 and group #2
  Other Names: Xylocaine
Drug: Triamcinolone Acetonide 40mg/mL — Transforaminal catheter-targeted ESI with triamcinolone acetonide 2 mL in group #2
  Other Names: Kenalog
  Arms: Transforaminal catheter-targeted ESI with triamcinolone

SUMMARY:
Do cervical epidural steroid injections done by transforaminal catheter targeted approach improve pain and function in patients with cervical radicular pain?

DETAILED DESCRIPTION:
Two distinct techniques used to administer epidural steroids specifically to the nerve root affected in a radicular pain syndrome, which include transforaminal access at the level of pathology and interlaminar interlaminar access at the C7-T1 level with subsequent advancement of an epidural cathether to the level of pathology. Use of an epidural catheter is necessary in order to achieve a targeted injection via an interlaminar approach in order to prevent dural puncture or direct spinal cord trauma. Anatomic studies confirm the distance between the ligamentum flavum and dura is on average, 4 mm at the C7-T1 or C6-C7 levels, but 1mm or smaller at C5-C6 and more rostral levels. Therefore, there is likely greater risk of dural puncture and spinal cord injury when "targeting" steroid delivery using only the interlaminar technique directly at the level where pathology is located (C4-C5, or C5-C6, for example). Thus, the interlaminar placement of a needle rostral to the C6-C7 level has been strongly discouraged.

Both the transforaminal injection approach and the targeted catheter approach demonstrate effectiveness. Studies have demonstrated the effectiveness of transforaminal epidural steroid injection for the treatment of cervical radicular pain. Our own recent work demonstrates the clinical effectiveness of the catheter-based targeted approach. However, these two approaches have never been directly compared. Thus, we aim to compare the differences in pain reduction, medication utilization, functional outcomes, patient satisfaction, and surgical rate reduction between these two approaches to the treatment of cervical radicular pain.

Cervical radicular pain is a common syndrome, often treated with epidural steroid injection (ESI). An approach that targets the therapeutic agent, corticosteroid, at the site of spinal pathology can be performed via a transforaminal approach or via a interlaminar approach at C7-T1 with subsequent epidural catheter advancement to the symptomatic level. There are no universal guidelines that recommend the use of one technique over the other. We will directly compare the clinical effectiveness of these two approaches as measured by pain reduction, medication utilization, functional outcomes, patient satisfaction, and surgical rate reduction. The results of this study will potentially influence clinical practice recommendations regarding the treatment of cervical radicular pain. If one technique proves superior, instating this technique will have implications potentially for reducing opioid use, surgery and other healthcare utilization, and general healthcare cost related to the treatment of cervical radicular pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80.
* Clinical diagnosis of unilateral C4-C8 radicular pain.
* Magnetic resonance imaging pathology consistent with clinical symptoms/signs.
* Numerical Rating Scale (NRS) pain score of 4 or higher.
* Pain duration of more than 6 weeks despite trial of conservative therapy (medications, physical therapy, or chiropractic care).

Exclusion Criteria:

* Refusal to participate, provide consent, or provide follow-up information for the 6-month duration of the study.
* Contraindications to Cervical Epidural Steroid Iinjection (CESI) (active infection, bleeding disorders, current anticoagulant or antiplatelet medication use, allergy to medications used for Cervical epidural steroid injection (CESI), and pregnancy).
* Cervical spinal cord lesions; cerebrovascular, demyelinating, or other neuro-muscular muscular disease.
* Current glucocorticoid use or Epidural Steroid Injection (ESI) within past 6 months.
* Prior cervical spine surgery.
* Patient request for or requirement of conscious sedation for the injection procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary L McCormick, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Radhakrishnan K, Litchy WJ, O'Fallon WM, Kurland LT. Epidemiology of cervical radiculopathy. A population-based study from Rochester, Minnesota, 1976 through 1990. Brain. 1994 Apr;117 ( Pt 2):325-35. doi: 10.1093/brain/117.2.325. PMID 8186959
- [Background] Carette S, Fehlings MG. Clinical practice. Cervical radiculopathy. N Engl J Med. 2005 Jul 28;353(4):392-9. doi: 10.1056/NEJMcp043887. No abstract available. PMID 16049211
- [Background] Heckmann JG, Lang CJ, Zobelein I, Laumer R, Druschky A, Neundorfer B. Herniated cervical intervertebral discs with radiculopathy: an outcome study of conservatively or surgically treated patients. J Spinal Disord. 1999 Oct;12(5):396-401. PMID 10549703
- [Background] Johnston MM, Jordan SE, Charles AC. Pain referral patterns of the C1 to C3 nerves: implications for headache disorders. Ann Neurol. 2013 Jul;74(1):145-8. doi: 10.1002/ana.23869. Epub 2013 Jun 17. PMID 23424170
- [Background] Mizutamari M, Sei A, Tokiyoshi A, Fujimoto T, Taniwaki T, Togami W, Mizuta H. Corresponding scapular pain with the nerve root involved in cervical radiculopathy. J Orthop Surg (Hong Kong). 2010 Dec;18(3):356-60. doi: 10.1177/230949901001800320. PMID 21187551
- [Background] Rhee JM, Yoon T, Riew KD. Cervical radiculopathy. J Am Acad Orthop Surg. 2007 Aug;15(8):486-94. doi: 10.5435/00124635-200708000-00005. PMID 17664368
- [Background] Malanga GA. The diagnosis and treatment of cervical radiculopathy. Med Sci Sports Exerc. 1997 Jul;29(7 Suppl):S236-45. doi: 10.1097/00005768-199707001-00006. PMID 9247921
- [Background] Renfrew DL, Moore TE, Kathol MH, el-Khoury GY, Lemke JH, Walker CW. Correct placement of epidural steroid injections: fluoroscopic guidance and contrast administration. AJNR Am J Neuroradiol. 1991 Sep-Oct;12(5):1003-7. PMID 1719788
- [Background] Mehta M, Salmon N. Extradural block. Confirmation of the injection site by X-ray monitoring. Anaesthesia. 1985 Oct;40(10):1009-12. doi: 10.1111/j.1365-2044.1985.tb10558.x. PMID 4061788
- [Background] Stojanovic MP, Vu TN, Caneris O, Slezak J, Cohen SP, Sang CN. The role of fluoroscopy in cervical epidural steroid injections: an analysis of contrast dispersal patterns. Spine (Phila Pa 1976). 2002 Mar 1;27(5):509-14. doi: 10.1097/00007632-200203010-00011. PMID 11880836
- [Background] Van Zundert J, Huntoon M, Patijn J, Lataster A, Mekhail N, van Kleef M; Pain Practice. 4. Cervical radicular pain. Pain Pract. 2010 Jan-Feb;10(1):1-17. doi: 10.1111/j.1533-2500.2009.00319.x. Epub 2009 Oct 5. PMID 19807874
- [Background] Johansson A, Hao J, Sjolund B. Local corticosteroid application blocks transmission in normal nociceptive C-fibres. Acta Anaesthesiol Scand. 1990 Jul;34(5):335-8. doi: 10.1111/j.1399-6576.1990.tb03097.x. PMID 2167604
- [Background] Benyamin RM, Singh V, Parr AT, Conn A, Diwan S, Abdi S. Systematic review of the effectiveness of cervical epidurals in the management of chronic neck pain. Pain Physician. 2009 Jan-Feb;12(1):137-57. PMID 19165300
- [Background] Stav A, Ovadia L, Sternberg A, Kaadan M, Weksler N. Cervical epidural steroid injection for cervicobrachialgia. Acta Anaesthesiol Scand. 1993 Aug;37(6):562-6. doi: 10.1111/j.1399-6576.1993.tb03765.x. PMID 8213020
- [Background] Castagnera L, Maurette P, Pointillart V, Vital JM, Erny P, Senegas J. Long-term results of cervical epidural steroid injection with and without morphine in chronic cervical radicular pain. Pain. 1994 Aug;58(2):239-243. doi: 10.1016/0304-3959(94)90204-6. PMID 7816491
- [Background] Saal JS, Saal JA, Yurth EF. Nonoperative management of herniated cervical intervertebral disc with radiculopathy. Spine (Phila Pa 1976). 1996 Aug 15;21(16):1877-83. doi: 10.1097/00007632-199608150-00008. PMID 8875719
- [Background] Riew KD, Yin Y, Gilula L, Bridwell KH, Lenke LG, Lauryssen C, Goette K. The effect of nerve-root injections on the need for operative treatment of lumbar radicular pain. A prospective, randomized, controlled, double-blind study. J Bone Joint Surg Am. 2000 Nov;82(11):1589-93. doi: 10.2106/00004623-200011000-00012. PMID 11097449
- [Background] Buttermann GR. Treatment of lumbar disc herniation: epidural steroid injection compared with discectomy. A prospective, randomized study. J Bone Joint Surg Am. 2004 Apr;86(4):670-9. PMID 15069129
- [Background] Huntoon MA. Anatomy of the cervical intervertebral foramina: vulnerable arteries and ischemic neurologic injuries after transforaminal epidural injections. Pain. 2005 Sep;117(1-2):104-11. doi: 10.1016/j.pain.2005.05.030. PMID 16055268
- [Background] Abbasi A, Malhotra G, Malanga G, Elovic EP, Kahn S. Complications of interlaminar cervical epidural steroid injections: a review of the literature. Spine (Phila Pa 1976). 2007 Sep 1;32(19):2144-51. doi: 10.1097/BRS.0b013e318145a360. PMID 17762818
- [Background] Rathmell JP, Benzon HT, Dreyfuss P, Huntoon M, Wallace M, Baker R, Riew KD, Rosenquist RW, Aprill C, Rost NS, Buvanendran A, Kreiner DS, Bogduk N, Fourney DR, Fraifeld E, Horn S, Stone J, Vorenkamp K, Lawler G, Summers J, Kloth D, O'Brien D Jr, Tutton S. Safeguards to prevent neurologic complications after epidural steroid injections: consensus opinions from a multidisciplinary working group and national organizations. Anesthesiology. 2015 May;122(5):974-84. doi: 10.1097/ALN.0000000000000614. PMID 25668411
- [Background] McCormick ZL, Nelson A, Bhave M, Zhukalin M, Kendall M, McCarthy RJ, Khan D, Nagpal G, Walega DR. A Prospective Randomized Comparative Trial of Targeted Steroid Injection Via Epidural Catheter Versus Standard C7-T1 Interlaminar Approach for the Treatment of Unilateral Cervical Radicular Pain. Reg Anesth Pain Med. 2017 Jan-Feb;42(1):82-89. doi: 10.1097/AAP.0000000000000521. PMID 27922950
- [Background] Ackerman WE 3rd, Ahmad M. The efficacy of lumbar epidural steroid injections in patients with lumbar disc herniations. Anesth Analg. 2007 May;104(5):1217-22, tables of contents. doi: 10.1213/01.ane.0000260307.16555.7f. PMID 17456677
- [Background] Gharibo CG, Varlotta GP, Rhame EE, Liu EC, Bendo JA, Perloff MD. Interlaminar versus transforaminal epidural steroids for the treatment of subacute lumbar radicular pain: a randomized, blinded, prospective outcome study. Pain Physician. 2011 Nov-Dec;14(6):499-511. PMID 22086091
- [Background] Schaufele MK, Hatch L, Jones W. Interlaminar versus transforaminal epidural injections for the treatment of symptomatic lumbar intervertebral disc herniations. Pain Physician. 2006 Oct;9(4):361-6. PMID 17066121
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Focus article: report of the NIH Task Force on Research Standards for Chronic Low Back Pain. Eur Spine J. 2014 Oct;23(10):2028-45. doi: 10.1007/s00586-014-3540-3. PMID 25212440
- [Background] Dworkin RH, Turk DC, McDermott MP, Peirce-Sandner S, Burke LB, Cowan P, Farrar JT, Hertz S, Raja SN, Rappaport BA, Rauschkolb C, Sampaio C. Interpreting the clinical importance of group differences in chronic pain clinical trials: IMMPACT recommendations. Pain. 2009 Dec;146(3):238-244. doi: 10.1016/j.pain.2009.08.019. PMID 19836888
- [Background] Kovacs FM, Abraira V, Royuela A, Corcoll J, Alegre L, Tomas M, Mir MA, Cano A, Muriel A, Zamora J, Del Real MT, Gestoso M, Mufraggi N; Spanish Back Pain Research Network. Minimum detectable and minimal clinically important changes for pain in patients with nonspecific neck pain. BMC Musculoskelet Disord. 2008 Apr 10;9:43. doi: 10.1186/1471-2474-9-43. PMID 18402665
- [Background] Gallizzi M, Gagnon C, Harden RN, Stanos S, Khan A. Medication Quantification Scale Version III: internal validation of detriment weights using a chronic pain population. Pain Pract. 2008 Jan-Feb;8(1):1-4. doi: 10.1111/j.1533-2500.2007.00163.x. PMID 18211588

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transforaminal ESI With Dexamethasone | Transforaminal Catheter-targeted ESI With Triamcinolone
Started | 60 | 60
Completed | 60 | 57
Not Completed | 0 | 3
Not completed — Did not receive allocated intervention. | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Interlaminar Catheter-targeted ESI With Triamcinolone: Group 2: Catheter-targeted cervical ESI with triamcinolone acetonide
  Transforaminal catheter-targeted ESI with triamcinolone: Catheter-targeted ESI via interlaminar access at the C7-T1 level with triamcinolone acetonide 2 mL (40mg/mL) and 1 ml 1% lidocaine (total volume 3 mL).
  Lidocaine: 1 mL of 1% lidocaine as diluent for the steroid in both group #1 and group #2
  Triamcinolone Acetonide 40mg/mL: Transforaminal catheter-targeted ESI with triamcinolone acetonide 2 mL in group #2
- Total: Total of all reporting groups
Arm/Group | Transforaminal ESI With Dexamethasone | Interlaminar Catheter-targeted ESI With Triamcinolone | Total
Number analyzed (Participants) | 60 | 57 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 48 | 99
  >=65 years | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 32 | 66
  Male | 26 | 25 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 60 | 57 | 117

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With Reduction of 50% or More of Neck and Arm Pain NRS Score
Description: The Percentage of Participants with Reduction of 50% or More of Neck and Arm Pain NRS score
Time Frame: 1 month follow up
Population: >50% Pain Reduction scored with 95% Confidence Interval.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transforaminal ESI With Dexamethasone | Interlaminar Catheter-targeted ESI With Triamcinolone
Number analyzed (Participants) | 60 | 57
percentage of participants | 49.1 [36.4 to 62.0] | 68.5 [54.9 to 79.5]

2. Secondary Outcome: Neck Disability Index-5
Description: Percentage of patients with >30% improvement in Neck Disability Index-5 score.
Time Frame: 1 month, 3 month, 6 month, and 1 year follow up
Population: Analysis was done for different timelines of one month, three months, six months, and one year.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transforaminal ESI With Dexamethasone | Transforaminal Catheter-targeted ESI With Triamcinolone
Number analyzed (Participants) | 60 | 57
percentage of participants
  One month | 48 [35 to 61] | 62 [49 to 75]
  Three month | 56 [43 to 69] | 58 [45 to 72]
  Six month | 55 [41 to 69] | 56 [43 to 69]
  One year | 47 [33 to 61] | 60 [47 to 74]

3. Secondary Outcome: Percentage of Participants Reporting >6.8 Reduction on the Medication Quantification Scale III
Description: The Medication Quantification Scale (MQS) is an instrument used for clinical and research applications for quantifying medication regimen use in chronic pain populations. A 6.8 point reduction is considered equivalent to 10 morphine eqivalents.
Time Frame: 1 month, 3 month, 6 month, and 1 year follow up
Population: Analysis was done for different timelines of one month, three months, six months, and one year.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transforaminal ESI With Dexamethasone | Transforaminal Catheter-targeted ESI With Triamcinolone
Number analyzed (Participants) | 60 | 57
percentage of participants
  One month | 16 [6 to 25] | 19 [8 to 29]
  Three month | 20 [9 to 31] | 17 [7 to 27]
  Six month | 15 [5 to 24] | 19 [8 to 29]
  One year | 7 [4 to 22] | 8 [6 to 27]

4. Secondary Outcome: The Percentage of Participants Reporting Patient Global Impression of Change Score of 6-7 (Indicating "Much Improved" and "Very Much Improved")
Description: Patient Global Impression of Change is a scale which measures participant reported satisfaction after an intervention. The outcome was measured as the percent of patients reporting a PGIC score of 6-7 (indicating "much improved" and "very much improved")
Time Frame: 1 month, 3 month, 6 month, and 1 year follow up
Population: Analysis was done for different timelines of one month, three months, six months, and one year.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Transforaminal ESI With Dexamethasone | Transforaminal Catheter-targeted ESI With Triamcinolone
Number analyzed (Participants) | 60 | 57
percentage of participants
  One month | 41 [28 to 54] | 59 [46 to 72]
  Three months | 42 [28 to 56] | 57 [43 to 70]
  Six months | 55 [40 to 69] | 53 [39 to 67]
  One year | 57 [42 to 73] | 61 [45 to 76]

ADVERSE EVENTS:
Time Frame: 1 year
Description: The definition does not differ from that outlined from clinicaltrials.gov
Arm/Group | Transforaminal ESI With Dexamethasone | Interlaminar Catheter-targeted ESI With Triamcinolone
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/57
Other Adverse Events (participants affected / at risk) | 0/60 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT03382821/Prot_SAP_000.pdf